CLINICAL TRIAL: NCT04590001
Title: A Feasibility Study Exploring the Effect of the MobiusHD® in Patients With Heart Failure
Brief Title: Effect of the MobiusHD® in Patients With Heart Failure
Acronym: HF-FIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD0593 0594 0595 0596 0610
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Mobius HD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MobiusHD (Experimental): Each subject enrolled in the study will undergo implantation of the MobiusHD device.
  Interventions: Device: MobiusHD

INTERVENTIONS:
Device: MobiusHD — The MobiusHD device is a nickel-titanium device that is implanted in the internal carotid sinus using a minimally invasive approach.

SUMMARY:
This is a prospective, multi-center, open-label clinical trial intended to evaluate the safety and effectiveness of the MobiusHD® in patients with heart failure and reduced ejection fraction.

DETAILED DESCRIPTION:
Subjects presenting with Class II, III or ambulatory IV heart failure with a left ventricular ejection fraction of ≤ 40% and NT-proBNP ≥ 400 will be considered for the study. Subjects who meet the initial screening requirements will undergo non-invasive imaging of the carotid anatomy to assess adequacy of the anatomy to allow placement of the MobiusHD device. Eligible subjects will receive an implant placed in the internal carotid artery.

Following implantation of the device, subjects will be seen at 1 week, 1, 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Currently NYHA Class II, III or ambulatory IV heart failure
3. Left ventricular ejection fraction ≤ 40%
4. NT-proBNP ≥ 400
5. Prescribed optimally-tolerated, stable, Guideline Directed Medical Therapy (GDMT) per country specific guidelines for the treatment of heart failure for at least 4 weeks
6. Six-minute hall walk (6MHW) distance of ≥ 150 m AND ≤ 400 m
7. Deemed an acceptable candidate for the implant procedure by the investigator

Exclusion Criteria:

1. Known or clinically suspected baroreflex failure or autonomic neuropathy
2. Currently implanted with a barostimulator device
3. Received cardiac resynchronization therapy (CRT) within six months of implantation
4. Received a CardioMEMS device within three months of the screening visit
5. History of any prior stroke with permanent neurologic defect or any prior intracranial bleed or other serious brain injury
6. Body mass index > 45
7. Serum estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
8. Presence of atherosclerotic plaque in the intended side for implantation as determined by carotid duplex
9. Internal ICA lumen diameters <5.0 mm or >11.75 mm within the planned location of the implant placement, or evidence of landing zone restrictions, such as inadequate length, vessel tapering, and/or vessel curvature that would preclude safe placement of the implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in New York Heart Association Heart Failure Class | 24 months
  Change in New York Heart Association Heart Failure Class between baseline and 3 months, 6 months, 12 months, 18 months and 24 months
Change in NT-proBNP blood test levels | 24 months
  Change in Amino-terminal prohormone of brain natriuretic peptide (NT-proBNP) between baseline and 3 months, 6 months, 12 months, 18 months, and 24 months
Change in QoL as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) and the EQ-5D Questionnaire. | 24 months
  Change in QoL measures between baseline and 3 months, 6 months, 12 months, 18 months, and 24 months will be measured. The KCCQ is used to measure the effect of heart failure on quality of life with a lower score indicating a worsening quality of life. The EQ-5D Questionnaire is a general measure of overall health with a lower score indicating a better overall health perception.
Change in 6MHW distance | 24 months
  Change in 6MHW distance between baseline and 3 months, 6 months, 12 months, 18 months and 24 months
Change in cardiac function / structure | 24 months
  Change will be evaluated using echocardiogram measured left ventricular ejection fraction, LV end diastolic volume, left atrial volume index, and severity of mitral regurgitation.
Adverse Events | 24 months
  Incidence and severity of adverse events and serious adverse events, including serious adverse cardiovascular and neurological events
Cardiovascular Mortality | 24 months
  Rate of cardiovascular mortality throughout the follow-up period will be reported.
Heart Failure Hospitalizations | 24 months
  Rate of heart failure hospitalizations throughout the follow-up period will be reported.

CONTACTS AND LOCATIONS:
Locations (17):
- Australia (2):
  - St. Vincent's Hospital, Darlinghurst, Sydney
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Canada (2):
  - London Health Science Center, London, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- Georgia (2):
  - Helsicore Ltd "Israeli-Georgian Medical Research Clinic Helsicore", Tbilisi
  - Tbilisi Heart and Vascular Center, Tbilisi
- Germany (7):
  - Charité Universitätsmedizin Berlin, Berlin
  - Heart Center, University Hospital Dresden, Dresden
  - CardioVascular Center - CVC Frankfurt, Frankfurt
  - Justus-Liebig-Universitat Giessen, Giessen
  - University of Saarlandes - Homburg, Homburg
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - University Hospital Ulm, Ulm
- Serbia (4):
  - Clinical Hospital Center Bežanijska Kosa, Belgrade, Belgrade
  - Institut for Cardiovascular Disease Dedinje, Belgrade, Belgrade
  - Institute for Cardiovascular Disease of Vojvodina, Kamenitz
  - University Clinical Center, Kragujevac, Kragujevac